CLINICAL TRIAL: NCT01371110
Title: Intravenous Ketamine in the Treatment of Obsessive-Compulsive Disorder
Acronym: IVKetamine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no funding
Sponsor: Wayne Goodman MD (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Wayne Goodman MD, Professor & Chair Psychiatry, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 11-1113; HSM#11-01536 (Other: THE MOUNT SINAI HEALTH SYSTEM)
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; Obsessive-Compulsive Disorder; ketamine; treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Active Comparator): Study participants will receive a one-time intravenous infusion of 0.5 mg/kg racemic ketamine hydrochloride
  Interventions: Drug: Ketamine
- Midazolam (Sham Comparator): Study participants will receive a one-time intravenous infusion of 0.045 mg/kg midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Ketamine hydrochloride is a nonbarbiturate anesthetic. It is formulated as a slight acid (pH 3.5 to 5.5) sterile solution for intravenous or intramuscular injection in concentrations containing the equivalent of either 50 or 100mg ketamine base per milliliter.
  Other Names: ketamine hydrochloride
  Arms: Ketamine
Drug: Midazolam — Midazolam is a short-acting benzodiazepine central nervous (CNS) depressant.
  Arms: Midazolam

SUMMARY:
Obsessive-Compulsive Disorder (OCD) is a chronic and disabling anxiety disorder and a leading cause of worldwide disability that presents a significant public health problem. Treatment options are limited and many OCD patients fail to respond completely or quickly to standard treatments, including pharmacotherapy and psychotherapy. At this time, patients who fail to respond to treatment with serotonergic drugs, augmenting antipsychotic agents, and behavioral therapy, have few additional treatment options aside from deep brain stimulation. Therefore, despite advances in current pharmacological and behavioral treatments, and the utility of serotonergic drugs, it is likely that other neurotransmitter systems are involved and that targeting these systems may increase treatment efficacy. Despite little evidence for serotonergic dysfunction in OCD, there is significant evidence that glutamatergic dysregulation may contribute to the development and progression of the disorder. Also, preliminary studies suggest that glutamatergic modulators (i.e. riluzole and d-cycloserine), particularly agents acting at the NMDA receptor (i.e. memantine), may be useful in OCD. The NMDA antagonist, ketamine, has demonstrated rapid effects when delivered as a single intravenous (IV) dose in depressed patients. Therefore, the objective of the current study is to investigate the safety and efficacy of a single dose of IV ketamine in treatment-resistant OCD.

DETAILED DESCRIPTION:
This study will test the safety and efficacy of a single intravenous (IV) dose of the N-methyl-D-aspartate (NMDA) glutamate receptor antagonist, ketamine, in treatment-resistant OCD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 21-65 years
* Women of childbearing potential must agree to use a medically accepted means of contraception for the duration of the study
* Primary diagnosis of Obsessive-Compulsive Disorder as assessed by the SCID-P, with symptoms for at least 1 year (Patients who meet criteria for OCD will be required to be medication free or have all psychotropics aside from SSRIs and as needed benzodiazepines tapered. Prior to study entry, proscribed psychotropics are tapered, and subjects must be on the same SSRI for at least 8 weeks with no change in dose for at least 4 weeks and throughout the study. However, subjects will be allowed to use benzodiazepines as needed throughout the study.)
* History of a failure to respond to at least two (2) adequate pharmacotherapy trials and CBT for OCD
* Subjects must have scored ≥ 21 on the Y-BOCS at Screening, and to not be in remission on Treatment Day #1, and Treatment Day #2
* Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document
* Subjects must be able to identify a family member, physician, or friend who will participate in the Treatment Contract and serve as an emergency contact.

Exclusion Criteria:

* Women who plan to become pregnant within the next six months, are pregnant or are breast-feeding
* Non-English speakers
* Any unstable medical illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG
* Lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, mental retardation, or pervasive developmental disorders
* Current evidence of psychotic or manic symptoms
* Drug or alcohol abuse or dependence within the preceding 6 months
* Lifetime abuse or dependence on ketamine or phencyclidine
* Patients judged by study investigator to be at high risk for suicide
* Current use of psychotropics other than SSRIs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne K Goodman, MD, Principal Investigator — Baylor College of Medicine (previously Icahn School of Medicine at Mount Sinai); Kyle Lapidus, MD, Principal Investigator — (previously Icahn School of Medicine at Mount Sinai)
Locations (1):
- Clinical Research Centers at Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mood and Anxiety Disorders Program (MAPs). In addition, referrals from clinicians in the Mount Sinai Medical Center, community clinics, and affiliated hospitals were also sought.
Pre-assignment Details: Eligible participants met treatment-resistant criteria if they failed to respond to ≥ 2 adequate pharmacotherapy trials with SRIs FDA approved medications for OCD with or without adjunctive antipsychotics, as well as cognitive behavioral therapy.
Groups:
- Ketamine (Randomized Week 1, Cross Over Midazolam Week 3)): Study participants will receive a one-time intravenous infusion of 0.5 mg/kg racemic ketamine hydrochloride
  Ketamine: Ketamine hydrochloride is a nonbarbiturate anesthetic. It is formulated as a slight acid (pH 3.5 to 5.5) sterile solution for intravenous or intramuscular injection in concentrations containing the equivalent of either 50 or 100mg ketamine base per milliliter.
- Midazolam (Randomized Wk 1, Cross Over Ketamine Wk 3): Study participants will receive a one-time intravenous infusion of 0.045 mg/kg midazolam
  Midazolam: Midazolam is a short-acting benzodiazepine central nervous (CNS) depressant.
Period: Overall Study
Arm/Group | Ketamine (Randomized Week 1, Cross Over Midazolam Week 3)) | Midazolam (Randomized Wk 1, Cross Over Ketamine Wk 3)
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine (Randomized Week 1, Cross Over Midazolam Week 3)) | Midazolam (Randomized Wk 1, Cross Over Ketamine Wk 3) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 49 [49 to 49] | 48.5 [34 to 63] | 48.6 [34 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCCS) Rating OCD Symptom Severity From Baseline to 24-hours After Ketamine Administration
Description: The primary efficacy outcome is change in the Y-BOCCS rating score on a scale from baseline to 24 hrs post-administration of ketamine.
  The 10 Y-BOCCS items are each scored on a four-point scale from 0 = "no symptoms" to 4 = "extreme symptoms." The sum of the first five items is a severity index for obsessions. The sum of the last five an index for compulsions. A translation of total score into an approximate index of overall severity is: 0-7 - subclinical; 8-15 - mild; 16-23 - moderate; 24-31 - severe; 32-40 - extreme.
Time Frame: Baseline and 24 Hours
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Ketamine (Randomized Week 1, Cross Over Midazolam Week 3)) | Midazolam (Randomized Wk 1, Cross Over Ketamine Wk 3)
Number analyzed (Participants) | 1 | 2
Units on a scale | -2.98 [-2.98 to -2.98] | -2.185 [-14.98 to 10.61]

2. Secondary Outcome: Percentage of Patients Who Meet Response and Remission
Description: Percentage of patients who meet response (defined as 25% reduction in Y-BOCCS score) and remission (defined as Y-BOCS score ≤10) criteria at 24 hrs post-infusion and durability of efficacy up to two weeks after administration. Assessments will be performed 24, 48 and 72 hrs post-infusion and after 7, 10, and 14 days.
Time Frame: up to 14 days
Measure: Number; unit: percentage of participants
Arm/Group | Ketamine (Randomized Week 1, Cross Over Midazolam Week 3)) | Midazolam (Randomized Wk 1, Cross Over Ketamine Wk 3)
Number analyzed (Participants) | 1 | 2
percentage of participants | 0 | 50

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=1) | Midazolam (N=2)
Suicidality (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to limited funding lead to small numbers of subjects analyzed (n=3) compared to what was planned (n=12).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No